CLINICAL TRIAL: NCT04128579
Title: A Phase 1b Multiple Ascending-dose Study of EQ001 in Subjects With Systemic Lupus Erythematosus With or Without Active Proliferative Lupus Nephritis
Brief Title: Study of EQ001 (Itolizumab) in Systemic Lupus Erythematosus With or Without Active Proliferative Nephritis
Acronym: EQUALISE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Equillium (Industry)
Collaborators: Biocon Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EQ001-19-002
Record Dates: First submitted 2019-09-30; First posted 2019-10-16 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Lupus Erythematosus; Lupus Nephritis
Keywords: Systemic Lupus Erythematosus; Active Proliferative Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — itolizumab

STUDY DESIGN:
Intervention Model Description: cohort based escalation of 6 subjects (Type A) single dose cohort of 20 subjects (Type B)
Masking Description: Type A and Type B are open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EQ001 Type A cohort (Experimental): EQ001 administered in an unblinded dose escalating cohort fashion by subcutaneous injection every two weeks for a total of 2 doses (up to 5 cohorts with dosing to be determined in the range of 0.4 -- 3.2 mg/kg).
  Interventions: Drug: Itolizumab [Bmab 600]
- EQ001 for Type B cohort (Experimental): EQ001 administered in an unblinded single dose cohort by subcutaneous injection every two weeks for a total of 13 doses (1.6 mg/kg).
  Interventions: Drug: Itolizumab [Bmab 600]

INTERVENTIONS:
Drug: Itolizumab [Bmab 600] — EQ001
  Other Names: Bmab600; Itolizumab

SUMMARY:
This is a multi-center study to evaluate the safety, tolerability, PK, PD, and clinical activity of itolizumab (EQ001) in subjects with Systemic Lupus Erythematosus with or without Active Proliferative Lupus Nephritis

DETAILED DESCRIPTION:
The study will enroll approximately 55 subjects, with up to 5 dose escalating cohorts of 6 open-label subjects enrolled for Type A-SLE and a single dose cohort of approximately 20 open-label subjects enrolled for Type B-Lupus Nephritis.

Subjects will receive itolizumab administered subcutaneously every two weeks for a total of either 2 (Type A) or 13 (Type B) doses with 4 or 12 weeks of follow-up after the last dose of investigational product.

ELIGIBILITY:
Type A Cohort Key Inclusion Criteria:

1. Is male or female, age ≥ 18 and ≤ 75 years
2. Has previously been documented to have met or currently meets Systemic Lupus International Collaborating Clinics (SLICC) and/or American College of Rheumatology (ACR) criteria for SLE
3. Received at least 1 immunosuppressive or immunomodulatory treatment for SLE at any time in the past or currently
4. Has documented elevation of antinuclear antibodies (ANA) in the past or during Screening
5. Restricted SLE treatments are stable and/or washed out
6. During Screening, has adequate hematologic function

Type B Cohort Key Inclusion Criteria:

1. Is male or female, age ≥ 18 and ≤ 75 years
2. Has a diagnosis of SLE
3. Kidney biopsy with a histologic diagnosis of LN Classes III or IV (+/- V)
4. Has a urine protein to creatinine ratio of > 1000 mg/g
5. Requires induction treatment due to newly diagnosed LN or relapsing/flaring disease or has an incomplete response to current treatment
6. Has adequate hematologic function
7. Restricted SLE treatments are stable and/or washed out
8. Most recent eGFR ≥ 40 mL/min/1.73m2
9. Has evidence of serologic activity

Key Exclusion Criteria:

1. Acute or chronic infections requiring systemic antibacterial, antifungal, or antiviral therapy
2. Positive for hepatitis B virus (HBV), hepatitis C virus (HCV), or HIV
3. Active TB or a positive TB test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2024-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kalunian, MD, Principal Investigator — UCSD
Locations (25):
- United States (19):
  - AKDHC Medical Research Services, LLC, Sun City, Arizona
  - California Institute of Renal Research, Chula Vista, California
  - University of California San Diego Perlman Ambulatory Clinic, La Jolla, California
  - Clinical Research of West Florida - Clearwater, Clearwater, Florida
  - Centre for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - University of Florida, Division of Rheumatology, Gainesville, Florida
  - Clinical Site Partners Leesburg, LLC, Leesburg, Florida
  - SouthCoast Research Center Inc, Miami, Florida
  - Hope Clinical Trials, Miami, Florida
  - Omega Research Maitland, LLC, Orlando, Florida
  - Clinical Research of West Florida - Tampa, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Georgia Nephrology, Lawrenceville, Georgia
  - Northwell Health / Division of Rheumatology, Great Neck, New York
  - Columbia University Medical Center, Div of Nephrology, New York, New York
  - Albert Einstein College of Medicine, Montefiore Medical Center, The Bronx, New York
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - Dallas Renal Group, Dallas, Texas
  - Prolato Clinical Research Center (PCRC), Houston, Texas
- India (4):
  - Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh
  - Medanta - The Medicity Hospital, Gurugramam
  - MAX Super Specialty Hospital, New Delhi
  - Jawaharlal Nehru Institute of Postgraduate Medical Education and Research (JIPMER), Puducherry
- Poland (2):
  - SP ZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi, Klinika Nefrologii, Hipertensjologii, Lodz
  - Miedzyleski Szpital Specjalistyczny w Warszawie, Oddzial Nefrologiczny i Stacja Dializ, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: company website — https://equilliumbio.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- EQ001 Type A Cohort (0.4mg/kg): EQ001 administered in an unblinded dose escalating cohort fashion by subcutaneous injection every two weeks for a total of 2 doses - 0.4mg/kg.
  Itolizumab [Bmab 600]: EQ001
- EQ001 Type A Cohort (0.8mg/kg): EQ001 administered in an unblinded dose escalating cohort fashion by subcutaneous injection every two weeks for a total of 2 doses - 0.8mg/kg.
  Itolizumab [Bmab 600]: EQ001
- EQ001 Type A Cohort (1.6mg/kg): EQ001 administered in an unblinded dose escalating cohort fashion by subcutaneous injection every two weeks for a total of 2 doses - 1.6mg/kg.
  Itolizumab [Bmab 600]: EQ001
- EQ001 Type A Cohort (2.4mg/kg): EQ001 administered in an unblinded dose escalating cohort fashion by subcutaneous injection every two weeks for a total of 2 doses - 2.4mg/kg.
  Itolizumab [Bmab 600]: EQ001
- EQ001 Type A Cohort (3.2mg/kg): EQ001 administered in an unblinded dose escalating cohort fashion by subcutaneous injection every two weeks for a total of 2 doses - 3.2mg/kg.
  Itolizumab [Bmab 600]: EQ001
Period: Overall Study
Arm/Group | EQ001 Type A Cohort (0.4mg/kg) | EQ001 for Type B Cohort | EQ001 Type A Cohort (0.8mg/kg) | EQ001 Type A Cohort (1.6mg/kg) | EQ001 Type A Cohort (2.4mg/kg) | EQ001 Type A Cohort (3.2mg/kg)
Started | 6 | 17 | 7 | 7 | 6 | 9
Completed | 6 | 14 | 6 | 6 | 5 | 4
Not Completed | 0 | 3 | 1 | 1 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EQ001 Type A Cohort (0.4mg/kg) | EQ001 for Type B Cohort | EQ001 Type A Cohort (0.8mg/kg) | EQ001 Type A Cohort (1.6mg/kg) | EQ001 Type A Cohort (2.4mg/kg) | EQ001 Type A Cohort (3.2mg/kg) | Total
Number analyzed (Participants) | 6 | 17 | 7 | 7 | 6 | 9 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (12.94) | 33.8 (11.18) | 44.6 (16.20) | 47.1 (6.82) | 48.2 (11.63) | 55.0 (11.09) | 45.3 (14.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 16 | 7 | 6 | 6 | 8 | 49
  Male | 0 | 1 | 0 | 1 | 0 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5 | 3 | 4 | 0 | 17
  Not Hispanic or Latino | 2 | 16 | 2 | 4 | 2 | 9 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 14 | 0 | 0 | 0 | 0 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 2 | 1 | 1 | 2 | 9
  White | 3 | 3 | 5 | 6 | 5 | 7 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 7 | 7 | 6 | 9 | 40
  India | 0 | 12 | 0 | 0 | 0 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events
Description: Number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Time Frame: Type A up to Day 57 or Type B up to Day 253
Measure: Count of Participants; unit: Participants
Arm/Group | EQ001 Type A Cohort (0.4mg/kg) | EQ001 for Type B Cohort | EQ001 Type A Cohort (0.8mg/kg) | EQ001 Type A Cohort (1.6mg/kg) | EQ001 Type A Cohort (2.4mg/kg) | EQ001 Type A Cohort (3.2mg/kg)
Number analyzed (Participants) | 6 | 17 | 7 | 7 | 6 | 9
Participants | 0 | 17 | 2 | 4 | 3 | 8

2. Secondary Outcome: To Characterize the PK of Itolizumab
Description: To characterize the pharmacokinetics of itolizumab
Time Frame: Type A up to Day 57 or Type B up to Day 253
Reporting Status: Not Posted

3. Secondary Outcome: CD6 Receptor Occupancy
Description: the % levels of free versus EQ001-bound CD6 receptor on T cells
Time Frame: Type A up to Day 57 or Type B up to Day 253
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The AEs that occurred after the first dose of itolizumab or during the study treatment and safety Follow-up Periods (Type A through Day 57; Type B through Day 253) were documented on the AE eCRF.
Arm/Group | EQ001 Type A Cohort (0.4mg/kg) | EQ001 for Type B Cohort | EQ001 Type A Cohort (0.8mg/kg) | EQ001 Type A Cohort (1.6mg/kg) | EQ001 Type A Cohort (2.4mg/kg) | EQ001 Type A Cohort (3.2mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/17 | 0/7 | 0/7 | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/17 | 0/7 | 0/7 | 0/6 | 1/9
Other Adverse Events (participants affected / at risk) | 0/6 | 17/17 | 2/7 | 4/7 | 3/6 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EQ001 Type A Cohort (0.4mg/kg) (N=6) | EQ001 for Type B Cohort (N=17) | EQ001 Type A Cohort (0.8mg/kg) (N=7) | EQ001 Type A Cohort (1.6mg/kg) (N=7) | EQ001 Type A Cohort (2.4mg/kg) (N=6) | EQ001 Type A Cohort (3.2mg/kg) (N=9)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Deterioration (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess on the proximal aspect of left thigh (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right elbow septic arthritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EQ001 Type A Cohort (0.4mg/kg) (N=6) | EQ001 for Type B Cohort (N=17) | EQ001 Type A Cohort (0.8mg/kg) (N=7) | EQ001 Type A Cohort (1.6mg/kg) (N=7) | EQ001 Type A Cohort (2.4mg/kg) (N=6) | EQ001 Type A Cohort (3.2mg/kg) (N=9)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 9 (9) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal ulceration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abcess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairement (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT04128579/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT04128579/SAP_001.pdf